CLINICAL TRIAL: NCT06873074
Title: Comparison of the Efficacy of Anterior and Posterior Long-segment Cervical Fixation for the Treatment of Lower Cervical Fractures in Ankylosing Spondylitis
Brief Title: A Retrospective Cohort Study About Surgical Efficacy for Lower Cervical Fractures in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Zhou Fang (Other)
Collaborators: Luohe Central Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Zhou Fang, Head of Orthopaedics, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: PekingUTH LXZ-AS
Record Dates: First submitted 2025-03-03; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ankylosing Spondylitis (AS); Spine Fracture
Keywords: Ankylosing Spondylitis; Cervical fracture and dislocation; anterior internal fixation and fusion; posterior internal fixation and fusion
MeSH Terms: conditions — Spondylitis, Ankylosing; Spinal Fractures; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- anterior group: anterior long segment cervical fixation
  Interventions: Procedure: anterior long segment cervical fixation
- posterior group: posterior long segment cervical fixation
  Interventions: Procedure: posterior long segment cervical fixation
- combined group: combined anterior and posterior fixation
  Interventions: Procedure: combined anterior and posterior fixation

INTERVENTIONS:
Procedure: anterior long segment cervical fixation
  Groups: anterior group
Procedure: posterior long segment cervical fixation
  Groups: posterior group
Procedure: combined anterior and posterior fixation
  Groups: combined group

SUMMARY:
The purpose of this retrospective cohort study was to observe and compare the efficacy of anterior cervical long segment fixation, posterior long segment fixation, and combined anterior and posterior fixation for the treatment of cervical vertebral fracture-dislocations in the lower cervical spine in ankylosing spondylitis.

DETAILED DESCRIPTION:
This was a retrospective cohort study. Patients operated for fracture-dislocation of the lower cervical vertebrae in ankylosing spondylitis in our hospital from 01/2014 to 01/2024 were retrospectively included as study subjects. Prior to the start of the study, an application will be made for approval through the hospital ethical committee, and the Declaration of Helsinki will be observed during the course of the study. The patients were divided into an anterior group (anterior long-segment cervical fixation), a posterior group (posterior long-segment cervical fixation), and a combined group (combined anterior and posterior fixation) according to the surgical access. The operation time, bleeding, complication occurrence, fracture healing and changes in neurological function of the three groups were compared. In this study, Frankel grading before and after surgery was used as the primary observation index, and operation time, intraoperative bleeding, occurrence of complications, and cervical fracture healing were used as the secondary observation index. SPSS 26.0 (IBM, New York, NY, USA) was applied for statistical analysis in this study.

ELIGIBILITY:
Inclusion criteria:

Meet the diagnostic criteria for ankylosing spondylitis, imaging showed that cervical ankylosing and fracture dislocation of the lower cervical vertebrae (cervical 3~7); Age 18~80 years old; undergo anterior, posterior or combined access internal fixation surgery and the fixation segment is ≥4 segments.

Exclusion criteria:

Systemic or local infection; Previous history of cervical vertebrae surgery; Postoperative loss of follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A multicenter-center retrospective cohort analysis of patients with ankylosing spondylitis (AS)-associated lower cervical fractures (C3-C7) treated between 2014 and 2023.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
complications | 1, 3, 6, and 12 months after the surgery at the final follow-up
  Categorized by the Clavien-Dindo classification system. Documented events include:
  Intraoperative: Dural tear, vertebral artery injury, nerve root injury.
  Postoperative (within 30 days): Surgical site infection, implant failure (screw loosening/breakage), cerebrospinal fluid leakage, dysphagia (anterior approach group), adjacent segment degeneration.
Radiographic Union Rate Assessed by X-ray and CT Criteria | 1, 2, 3, 6, and 12 months after the surgery at the final follow-up
  X-ray union: Fracture line blurring with callus formation ≥50% of fracture area on anteroposterior/lateral views.
  CT union: Complete fracture line disappearance with continuous callus bridging on thin-slice (≤1 mm) CT reconstructions.
Frankel Grade Improvement Rate and Neurological Recovery Index | 1, 3, 6, and 12 months after the surgery at the final follow-up
  Assessment tool: Frankel Spinal Cord Injury Scale (A: complete paralysis; B: sensory preservation only; C: non-functional motor preservation; D: functional motor preservation; E: normal function).
  Improvement rate: Defined as ≥1-grade improvement from baseline, reported as frequency (percentage).
  Recovery index: Calculated by assigning numerical values (A=1 to E=5), with differences between preoperative and final grades expressed as mean ± SD.
  Severe injury recovery: Proportion of patients with preoperative Frankel B/C grades achieving D/E grades postoperatively.

SECONDARY OUTCOMES:
Operative time | immediately after surgery
  Defined as the duration from skin incision to wound closure (minutes). Data will be presented as mean ± standard deviation (SD) and compared among anterior, posterior, and combined approach groups.
Intraoperative blood loss: | immediately after surgery
  Calculated using suction drainage volume combined with gauze weight measurement (1 g ≈ 1 mL). Reported as median (range) and mean ± SD.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No